CLINICAL TRIAL: NCT04784195
Title: Functional and Morphological Characteristics of Neck Muscles in Acrobatic Skydivers: an Observational Prospective Cohort Study
Brief Title: Functional and Morphological Characteristics of Neck Muscles in Acrobatic Skydivers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Javier Reina Abellan, Director, Universidad de Murcia
Other Study IDs: CE102001
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Neck Muscle Issue; Sternocleidomastoid; Contracture; Deltoid Muscle Strain
MeSH Terms: conditions — Congenital torticollis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Profesional acrobatics: Profesional Acrobatic Skyedivers as the cort group
  Interventions: Behavioral: Observation
- General active participations: Adults with meched caracteristics with the profesional acrobatics

INTERVENTIONS:
Behavioral: Observation — Verification of morfology and functionality of neck muscles
  Groups: Profesional acrobatics

SUMMARY:
An observational cohort study, following the Strengthening the Reporting of Observational Studies in Epidemiology(STROBE) guidelines.

Two groups will be examined, a group composed by spanish acrobatic skydivers and a control group composed by general physically active population(GPAP).

DETAILED DESCRIPTION:
Two groups will be examined for veryfing the morfology and the function of neck muscles.

The profesional group composed by spanish acrobatic skydivers and a general group composed by general physically active population(GPAP). Both groups are matched at known confounder outcomes such as: physical activity level, age, sex, body weight and history of neck pain. Frequency matching will be carried out, subjects will be matched on known confounders.

ELIGIBILITY:
Inclusion Criteria:

* pain-free in the neck area in the last three months
* didn't actually take any drugs that can interfere with muscle strength

Exclusion Criteria:

* participants that not mached with the skydivers caracteristics

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants with a high level of physical activity and actualy involved in skydiving practices.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Anticipatory postural adjustment | 10 minutes
  Electromyographic test in ms.The myoelectric signal will be recorded by using mDurance R system (mDurance Solutions SL, Granada). The electrodes used will be pre-gelled Ag/AgCl with a diameter of 10mm and an interelectrode distance of 20mm.
Isometric cervical strength | 10 minutes
  Measured in newton with heandheld Dynamometer (model 001165, Lafayette Instrument Company)
Neck flexor and extensor endurance | 10 minutes
  Measures in seconds with a stopwatch